CLINICAL TRIAL: NCT01151267
Title: Hypercapnic Spontaneous Hyperpnoea and Recovery From Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHN REB 08-0017-B
Record Dates: First submitted 2010-05-17; First posted 2010-06-28 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Anesthesia; Surgery
Keywords: Isocapnic hyperpnoea (IH); Anesthesia; Accelerate elimination of inhalation agents; Recovery from anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Other): The O2 flow on the anesthetic machine will be set at 15 L/min. Ventilatory assistance will be performed to maintain O2 saturation >97% and end tidal CO2 at 35-45mmHg.
  Interventions: Other: Standard Anesthesia management for post surgical patients
- HSH Group (Active Comparator): Patient will be disconnected from the anesthetic circuit and connected to the resuscitation bag attached to the IH system. With O2 flow of 2 L/min patient will be gently ventilated until recovery of the spontaneous ventilation. After starting spontaneous ventilation basal O2 flow will be adjusted to keep ETCO2 in range of 50-60 mm Hg or minute ventilation of 15-17 L/min, whichever occurs first.
  Interventions: Device: Hypercarbic Spontaneous Hyperpnoea

INTERVENTIONS:
Other: Standard Anesthesia management for post surgical patients — The O2 flow on the anesthetic machine will be set at 15 L/min. Ventilatory assistance will be performed to maintain O2 saturation >97% and end tidal CO2 at 35-45mmHg.
  Arms: Control Arm
Device: Hypercarbic Spontaneous Hyperpnoea — Patient will be disconnected from the anesthetic circuit and connected to the resuscitation bag attached to the IH system. With O2 flow of 2 L/min patient will be gently ventilated until recovery of the spontaneous ventilation. After starting spontaneous ventilation basal O2 flow will be adjusted to keep ETCO2 in range of 50-60 mm Hg or minute ventilation of 15-17 L/min, whichever occurs first.
  Arms: HSH Group

SUMMARY:
The rate of elimination of inhalation agent is directly proportional to the degree of alveolar ventilation. Using Isocapnic Hyperpnoea (IH) device, it is possible to maintain constant end-tidal CO2 with increased minute ventilation. This is achieved by passively adding a flow of CO2 to the inspirate in proportion to increases in ventilation above the baseline. In animal and human studies IH shortens the time of awakening from isoflurane and sevoflurane anesthesia when manual positive pressure ventilation is applied. IH device could be used for spontaneous hyperpnoea as well. The investigators want to compare recovery times from sevoflurane anesthesia in patients with application of hypercapnic spontaneous hyperpnoea (HSH) versus the standard anesthesia protocol (controls). 44 patients ill be randomized to either HSH facilitated recovery, or conventional recovery (controls).The time intervals from the end of anesthesia (turning off the vaporizer) until recovery milestones will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* elective gynecological surgery
* age 18-80
* ASA I-III
* informed consent

Exclusion Criteria:

* ASA IV-V,
* contra-indications to sevoflurane anesthesia or other anesthetics included in the protocol
* history of cardiac or respiratory disease
* intracranial pathology
* alcohol or drug abuse
* psychiatric illness and/or medications

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time from the end of anesthesia to the readiness for post-anesthesia care unit (PACU) discharge. | End of anesthesia (turning off the vaporizer) until readiness for PACU discharge, approximately 30 minutes to 2 hours

SECONDARY OUTCOMES:
Comparison of pain and sedation scores | End of anesthesia (turning off the vaporizer) to PACU discharge, approximately 30 minutes to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada